CLINICAL TRIAL: NCT03926923
Title: Analysis of Mother-child Interaction as Well as Expression and Methylation of Candidate Genes of Stress Signaling Pathways in Mature Infants
Brief Title: Analysis of Mother-child Interaction and Regulation of Candidate Genes of Stress Signaling Pathways in Mature Infants
Status: Completed | Type: Observational
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Katrin Mehler, adjunct professor, medical doctor Katrin Mehler, University of Cologne
Other Study IDs: 19-1118
Record Dates: First submitted 2019-04-02; First posted 2019-04-25 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Mother-Child Interaction
Keywords: stress response; neurodevelopment; newborn
MeSH Terms: conditions — Fractures, Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * 500µl whole blood sample for RNA extraction in peripheral white blood cells
  * 2 buccal swabs with mucosal epithelial cells for RNA and DNA extraction
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — There will be no intervention. The blood sample is taken while a routine blood sampling.

SUMMARY:
The planned study will investigate the quality of mother-child interaction at the age of 6 months as well as the expression and methylation of candidate genes of stress signaling pathway in mature infants.

At best, mother and the healthy, term newborn are undisturbed after birth. This creates optimal conditions for the development of a good mother-child interaction. The results of the mother-child interaction and the molecular genetic investigations will be compared to the results of the randomized controlled delivery room skin-to-skin study (deisy, clinicaltrial.gov identifier: NCT 01959737). This study showed a significant difference in the mother-child interaction and expression of candidate genes in preterm infants with or without skin-to-skin contact after birth.

The investigators hypothesize that the quality of mother-child interaction at the age of six months will be better in term newborns without postpartal separation of mother and child than in preterm infants with or without skin contact after birth. The second hypothesis is that there will be a difference in the expression and methylation of candidate genes of stress signaling pathway in these infants.

DETAILED DESCRIPTION:
A separation of mother and child after birth can influence the quality of mother-child interaction and the regulation of stress signaling pathways. Maternal depression, parental stress and socioeconomic status can also affect the quality of mother-child interaction.

A former controlled randomized delivery room skin-to-skin study (deisy) showed, that skin contact of preterm infants and their mothers after birth improves the mother-child interaction. It also leads to a differential expression of candidate genes of the stress signaling pathways, which suggests a long term effect on mechanisms in stress response. The study group should now be compared to a group of mature infants with a normal, uninterrupted postnatal course.

The hypothesis is that the intervention in the deisy study (early skin-to-skin contact of preterm infants and their mothers) improves the mother-child interaction so that it is nearly comparable to mature infants with uninterrupted mother-child contact after birth. Furthermore it is assumed that the expression and methylation of candidate genes of the stress signaling pathways will be influenced by the intervention in the same way.

The mother-child interaction will be evaluated at the age of six months with a standardized method (Mannheim Rating Scales). Questionnaires about maternal depression, social support, socio-economic status, parental stress and mother-child relationship disorders as well as samples for the molecular genetic testing will be collected on the third day of life and at the age of six months. For the molecular genetic testing one blood sample and buccal swabs will be taken. The blood sample will not be done additionally but with a routine blood sampling on the third day of life (screening of inborn errors of metabolism).

ELIGIBILITY:
Inclusion Criteria:

* mature newborn (38 to 41 weeks of gestational age)
* first child
* no separation of mother and child for three hours after birth
* informed consent

Exclusion Criteria:

* multiples
* malformations or syndromes in the infant
* maternal psychological or severe physical illness

Ages: 1 Day to 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population consits of healthy mature newborns who are not seperated from the mothers for three hours after birth. The recruitment will take place in three obstetric hospitals in Cologne (University Hospital of Cologne, Krankenhaus der Augustinnerinnen, evangelisches Krankenhaus Köln-Weyertal).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-07-18 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Analysis of the mother-child interaction of mature infants at the age of six months | at the age of six months
  Mother-child interaction is investigated at the age of six months using Mannheim Rating Scales. Therefore a four-minute-videotape of the mother changing the infant's diapers and playing with the infant is used.
  Mannheim Rating Scales is a good validated standardized observation instrument. Stimulation and response from the mother as well from the infant are being recorded. Different communication channels can be used by mother and child (vocal, facial or motor).
  All behaviors are analysed at intervals of five seconds (event coding). Then the values are formed from the sum of the coded events.
  The scale ranges from 0 to 48. If there is no interaction, the scale is 0. If there is an interaction in each interval (every 5 seconds in a 4 minute videotape), the scale is 48. The mother-child interaction is better if the scale is higher.

SECONDARY OUTCOMES:
Analysis of expression and methylation of candidate genes of stress signaling pathways from infant blood (on the third day of life) as well as mucosal epithelial cells (buccal swab on the third day of life and at the age of six months) | third day of life and age of six months
  RNA and DNA will be extracted from peripheral white blood cells and mucosal epithelial cells. The expression and methylation of candidate genes of the stress signaling pathways are investigated. The candidate genes are glucocorticoid receptor (NR3C1), corticotropin releasing hormone (CRH), corticotropin-releasing hormone receptor 1 (CRHR1), serotonin receptors (1A and 2A), serotonin transporter (slc6a4) and vasopressin.
Maternal depression | third day of life and age of six months
  Maternal depression is assessed with the German long form of the Center for Epidemiological Studies Depression Scale (CES-D). It is a self-report questionnaire to measure depressive symptoms and it consists of 20 questions. For each question the response choice are assigned point values (how often a symptom occurred during the last week). The point values are summed to a total measure score. The score ranges from 0 to 60. Zero points represents no symptoms of depression, a score of 15 or higher is interpreted to indicate a risk of depression.
Social support | third day of life and age of six months
  Social support is assessed with the short version of the F-SozU (Fragebogen zur sozialen Unterstützung, questionnaire on social support) scale (F-SozU K-22).
  The questionnaire records the subjectively perceived or anticipated support from the social environment. There are 22 items and the test person can indicate the degree of agreement on a five-level Likert scale (from 1 = does not apply to 5 = applies completely). The scale ranges from a minimum of 22 points to a maximum of 110 points. The higher the score, the better the subjectively perceived or anticipated support.
socio-economic status | third day of life and age of six months
  There will be a question to the household income per month and the mother's highest school-leaving certificate.
parental stress | third day of life and age of six months
  Parental stress is assessed with the German form of the parenting stress index (PSI).
  It consists of 48 items. The test person can indicate the degree of agreement on a five-level Likert scale (from 1 = does not apply to 5 = applies completely). There are 12 subscales, each consisting of 4 items and the points on the Likert scale are added. In each subscale there can be a minimum of 4 and a maximum of 20 points. The higher the score, the higher the parental stress.
Parental Bonding | third day of life and age of six months
  Parental Bonding is assessed with the parental bonding questionnaire (PBQ). It consists of 25 items and each item is rated on a scale from 0 to 3 points (response range from "very like" to "very unlike"). There are four subscales and the point values of each subscale are summed to a total measure score. The four subscales are: impaired bonding, rejection and anger, anxiety about care, risk of abuse. The higher the score, the higher the risk of a disorder in each area of the subscale.

CONTACTS AND LOCATIONS:
Overall Officials: Katrin Mehler, MD, Principal Investigator — University of Cologne
Locations (1):
- University hospital of Cologne, Department of Neonatology, Cologne, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mehler, K.; Hucklenbruch-Rother, E.; Trautmann-Villalba, P.; Keller, T.; Becker, I.; Kribs, A. (2018): Early skin-to-skin contact in preterm infants is safe and improves quality of mother-child interaction. Abstracts der 44. Jahrestagung der Gesellschaft für Neonatologie und Pädiatrische Intensivmedizin (GNPI) In: Monatsschr Kinderheilkd (166), S. S54.
- [Background] Hucklenbruch-Rother, E.; Mehler, K.; Keller, T.; Vohlen, C.; Mehdiani, N.; Kribs, A. (2018): Early skin-to-skin-contact affects stress response gene expression at hospital discharge. Abstracts der 44. Jahrestagung der Gesellschaft für Neonatologie und Pädiatrische Intensivmedizin (GNPI) In: Monatsschr Kinderheilkd (166), S. S54-S55
- See also: deisy study results - improvement of mother-child interaction — https://doi.org/10.1007/s00112-018-0501-7
- See also: deisy study results - effect on stress response gene expression — https://doi.org/10.1007/s00112-018-0501-7